CLINICAL TRIAL: NCT01892631
Title: A Feasibility Study for a Cluster Randomised Trial of Text Messaging Reminders for Influenza Vaccine in Patients Under 65 in Clinical Risk Groups in English Primary Care.
Brief Title: Text Messaging Reminders for Influenza Vaccine in Primary Care
Acronym: TXT4FLUJAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: txt4flujab
Record Dates: First submitted 2013-06-13; First posted 2013-07-04 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: Text messaging
MeSH Terms: conditions — Influenza, Human | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Other): Practices in the standard care arm will proceed with their seasonal influenza campaign as planned.
  Interventions: Other: Standard care
- Text messaging intervention (Experimental): Practices in the text messaging intervention arm will be asked to send a text message to patients under 65 at risk of influenza.
  Interventions: Other: Text message influenza vaccination reminder

INTERVENTIONS:
Other: Text message influenza vaccination reminder — Practices in the text messaging intervention arm will be asked to send a text message to patients under 65 at risk of influenza.
  Arms: Text messaging intervention
Other: Standard care — Practices in the standard care arm will be asked to proceed with their seasonal influenza campaign as planned.
  Arms: Standard care

SUMMARY:
Influenza morbidity and mortality cause a substantial financial burden to the NHS and to the UK as a whole. Influenza vaccine is safe and effective but is required annually because the circulating strain of virus changes each year. In the UK in 2012, the Chief Medical Officer (CMO) recommended that at least 75% of elderly people (aged 65+) and 75% people under 65 with certain chronic conditions (e.g. chronic heart disease, diabetes, asthma, etc) should be vaccinated. While primary care practices are achieving these targets for elderly patients, those set for younger patients with chronic conditions are not being met, with a third of patients being missed in the 2011/12 flu season and with no substantial improvements in uptake in the past decade. Therefore strategies to increase flu vaccine uptake in these patients are required.

Previous trials have shown that patient reminders can increase vaccine uptake and in particular, text messaging has shown to work in some populations in the United States as a cheap, simple and effective reminder. However, whether the same is true in UK general practice is unclear. The use of text messaging in the NHS for appointment reminders is also increasing as it is cheap, quick and effective. Text messaging is already used in roughly 30% of practices to remind patients about their flu vaccine but there has been no trial addressing its effectiveness. Therefore, we propose a trial of a text messaging flu vaccine reminder in patients aged under 65 who have a chronic condition. We hypothesise that practices that send a text message will have increased flu vaccine uptake.

ELIGIBILITY:
Inclusion Criteria:

* practices must use text messaging software to communicate with patients;
* practices must not have used a text message to remind patients aged under 65 about influenza vaccine in the 2012/13 influenza season.
* practices will send the text message to eligible patients who are aged between 18 and 65, with one of the following risk conditions: chronic respiratory disease, chronic liver disease, chronic kidney disease, chronic heart disease, chronic neurological disease, immunosuppression

Exclusion Criteria:

* practices will not send the text message to pregnant women.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients at risk who received flu vaccine | up to 9 months

SECONDARY OUTCOMES:
Proportion of practices reporting 'yes' to difficulties | up to 3 months
  Proportion of practices reporting 'yes' that they had difficulties in sending the text message to patients
Recruitment rate | 3 months after initial contact
  This is a pilot feasibility study and recruitment of practices to the trial is an outcome.
Practice delivery of text message | One month after study start (October 1st 2013)
  Did the practice send the text message to eligible patients and was the content of the message as described in the protocol.
Were outcome data available | up to 9 months
  Were outcome data regarding text message and flu vaccine uptake available.

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Hygiene and Tropical Medicine, London, Select County, United Kingdom